CLINICAL TRIAL: NCT06996886
Title: An Open-Label, Randomized, Four-Treatment, Four-Period, Single-Dose Crossover Study in Healthy Participants to Assess the Relative Bioavailability of AZD5004 in Three Solid Oral Formulations (F1, F3, F4)
Brief Title: A Study in Healthy Participants to Investigate Relative Bioavailability of AZD5004 in Three Solid Oral Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7260C00012
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: Relative bioavailability; GLP-1 receptor agonist; Type 2 Diabetes Mellitus; Obesity; Oral tablet formulations
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence A (Experimental): Participants will receive single dose of AZD5004 on Day 1 in F1 (fasted) (Treatment period 1), on Day 8 in F4 (fasted) (Treatment period 2), on Day 15 in F4(fed) (Treatment Period 3) followed by on Day 22 in F3 (fasted) (Treatment Period 4) respectively.
  Interventions: Drug: AZD5004
- Treatment Sequence B (Experimental): Partcipants will receive single dose of AZD5004 on Day 1 in F4 (fasted) (Treatment Period 1), on Day 8 in F4 (fed) (Treatment Period 2), on Day 15 in F3 (fasted) (Treatment Period 3) followed by on Day 22 in F1 (fasted) (Treatment Period 4) respectively.
  Interventions: Drug: AZD5004
- Treatment Sequence C (Experimental): Participants will receive single dose of AZD5004 on Day 1 in F4 (fed) (Treatment Period 1), on Day 8 in F3 (fasted) (Treatment Period 2, on Day 15 in F1 (fasted) (Treatment Period 3 followed by on Day 22 in F4 (fasted) (Treatment Period 4) respectively.
  Interventions: Drug: AZD5004
- Treatment Sequence D (Experimental): Participants will receive single dose of AZD5004 on Day 1 in F3 (fasted) (Treatment Period 1), Day 8 in F1 (fasted) (Treatment Period 2), on Day 15 in F4 (fasted) (Treatment Period 3) followed by Day 22 in F4 (fed) (Treatment Period 4) respectively.
  Interventions: Drug: AZD5004

INTERVENTIONS:
Drug: AZD5004 — Participants will be receiving three different formulations (F1, F3, and F4) as single dose of AZD5004 orally in fasted and fed state.

SUMMARY:
The purpose of this study is to assess the relative bioavailability of a single dose AZD5004 in healthy participants, among 3 different oral tablet formulations.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, 4-period, 4-treatment, single-dose crossover study in healthy participants.

Participants will receive one single dose of AZD5004 at the beginning of each of the four Treatment Periods, and a total of 4 doses of AZD5004. Three different formulations (F1, F3, and F4) will be used across the Treatment Periods.

The study comprises of total four treatment periods.

* A Screening Period of maximum 27 days. Four Treatment Periods of 7 days each.
* Treatment Period 1 (Day -1 to Day 6)
* Treatment Period 2 (Day 7 to Day 13)
* Treatment Period 3 (Day 14 to Day 20)
* Treatment Period 4 (Day 21 to Day 27)
* A final Follow-up Visit within 7 to 10 days after the last study intervention administration (Day 22 of Treatment Period 4).

The treatments are as follows:

* Treatment 1: Single dose of AZD5004 in Formulation 1 (F1) -fasted
* Treatment 2: Single dose of AZD5004 in Formulation 4 (F4) -fasted
* Treatment 3: Single dose of AZD5004 in F4- fed
* Treatment 4: Single dose of AZD5004 in Formulation 3 (F3) - fasted

Participants will be randomized equally to one of the following treatment sequences:

* Treatment Sequence A: F1, F4, F4 (fed), F3
* Treatment Sequence B: F4, F4 (fed), F3, F1
* Treatment Sequence C: F4 (fed), F3, F1, F4
* Treatment Sequence D: F3, F1, F4, F4 (fed)

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy male and female participants with suitable veins for cannulation or repeated venipuncture.
* Female participants:

  1. Female(s) of childbearing potential: If heterosexually active must agree to use an approved method of highly effective contraception.
  2. Female(s) not of childbearing potential
* Male participants:

  1. Condom use is required for the duration of the clinical study.
  2. Additional contraception must be used for the sexual partners of male study participants throughout the clinical study.
* Have a Body Mass Index (BMI) ≥ 23 kg/m2 and not exceeding 35 kg/m2 inclusive (at the time of Screening) and weigh at least 60 kg.

Main Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study
* History of acute pancreatitis (unless due to previously resolved gallstone pancreatitis and post-cholecystectomy), chronic pancreatitis, gallstones, or elevation in serum lipase/pancreatic amylase.
* Clinically significant inflammatory bowel disease, gastroparesis, severe disease, or surgery affecting the upper GI tract (including bariatric surgery).
* Any clinically important illness, medical/surgical procedure, or trauma.
* Any laboratory values with the deviations specified in protocol and clinically important abnormalities in clinical chemistry, hematology, or urinalysis results.
* Any positive result at Screening for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb) or Human immunodeficiency Virus (HIV).
* Abnormal vital signs, after 10 minutes supine rest, at Screening and/or admission to the Clinical Unit.
* Serum triglyceride concentrations above 1000 mg/dL (11 mmol/L).
* Basal calcitonin level > 50 ng/L or pg/mL at Screening or history/family history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia (MEN), type 2.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol
* Positive screen for drugs of abuse, or alcohol or cotinine (nicotine).
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5004.
* Excessive intake of caffeine-containing drinks or food
* History of psychosis or bipolar disorder and major depressive disorder.
* History of suicide attempt or history of suicidal ideation within the past year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the relative bioavailability of AZD5004 in 3 different solid oral formulations (F1, F3, F4)
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the relative bioavailability of AZD5004 in 3 different solid oral formulations (F1, F3, F4)
Maximum observed drug concentration (Cmax) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the relative bioavailability of AZD5004 in 3 different solid oral formulations (F1, F3, F4)
Time to reach maximum observed concentration (tmax) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the relative bioavailability of AZD5004 in 3 different solid oral formulations (F1, F3, F4)
Half-life (t½) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the relative bioavailability of AZD5004 in 3 different solid oral formulations (F1, F3, F4)
Apparent total body clearance (CL/F) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the relative bioavailability of AZD5004 in 3 different solid oral formulations (F1, F3, F4)

SECONDARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the food effect on the relative bioavailability of AZD5004 in one solid oral formulation (F4)
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the food effect on the relative bioavailability of AZD5004 in one solid oral formulation (F4)
Maximum observed drug concentration (Cmax) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the food effect on the relative bioavailability of AZD5004 in one solid oral formulation (F4)
Time to reach maximum observed concentration (tmax) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the food effect on the relative bioavailability of AZD5004 in one solid oral formulation (F4)
Half-life (t½) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the food effect on the relative bioavailability of AZD5004 in one solid oral formulation (F4)
Apparent total body clearance (CL/F) | Day 1-6, Day 8-13, Day 15-20 and Day 22-27
  To assess the food effect on the relative bioavailability of AZD5004 in one solid oral formulation (F4)
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Screening (Day -28 to Day -2) up to Follow-up (Day 29 to Day 32)
  To study the safety and tolerability of a single dose AZD5004 in 3 different solid oral formulations (F1, F3, F4), and F4 under fasted and fed conditions in healthy participants

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/